CLINICAL TRIAL: NCT02679807
Title: Effect of Probiotic on Rhinovirus Induced Colds
Acronym: MK EPRIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Danisco Sweeteners Oy (Industry)
Responsible Party: Principal Investigator, Ronald Turner, MD, Professor, Department of Pediatrics, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 18625
Record Dates: First submitted 2016-02-08; First posted 2016-02-10 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold | interventions — Sucrose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bifidobacterium lactis Bl-04 (Active Comparator): 2*109 cfus of probiotic Bifidobacterium lactis Bl-04 (DuPont Nutrition and Health) mixed with 1g of sucrose as a carrier
  Interventions: Biological: Bifidobacterium animalis subsp. lactis Bl-04
- Placebo (Placebo Comparator): sucrose
  Interventions: Other: sucrose

INTERVENTIONS:
Biological: Bifidobacterium animalis subsp. lactis Bl-04
  Arms: Bifidobacterium lactis Bl-04
Other: sucrose
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind placebo controlled trial to evaluate the effect of a probiotic (Bl-04) on the occurrence of rhinovirus-associated common cold illness in the experimental rhinovirus challenge model. A previous study documented that Bl-04 has significant effects on the innate immune response in the nose and this study will be powered to assess whether these effects translate into a demonstrable clinical benefit. Volunteers will be given Bl-04 or placebo for 28 days then challenged with rhinovirus. The primary analysis will be on the proportion of volunteers who develop a rhinovirus associated illness in the two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA AT ENROLLMENT:

* Subject must be 18-60 years of age.
* Subject must read and sign a copy of the approved Consent Form
* Subject must have a serum neutralizing antibody titer of less than or equal to 1:4 to rhinovirus type 39

INCLUSION CRITERIA AT DAY -28

• Female subjects must be using an effective birth control method.

INCLUSION CRITERIA AT CHALLENGE:

* Female subjects must be using an effective birth control method.

Exclusion Criteria:

* Antibiotic use within 3 months prior to day -28

  * Female subjects with a positive urine pregnancy screen
  * History of use of probiotics in the preceding two weeks
  * Current cancer diagnosis or immunosuppressive therapy in the last 6 months
  * Any clinically significant abnormalities of the upper respiratory tract
  * Any clinically significant acute or chronic respiratory illness
  * Any clinically significant bleeding tendency by history
  * Hypertension that requires treatment with antihypertensive medications
  * History of angina or other clinically significant cardiac disease
  * Any medical condition that in the opinion of the Principal Investigator is cause for exclusion from the study
  * History of regular use (more than 3 days in 7) of tobacco products within the preceding two weeks
  * History of drug or alcohol abuse in the 6 months preceding the study

EXCLUSION CRITERIA AT CHALLENGE:

* Any upper respiratory infection or allergic rhinitis in the two weeks prior to the challenge
* Female subjects with positive pregnancy screen prior to challenge
* Any medical condition that in the opinion of the Principal Investigator is cause for exclusion from the study
* Use of any anti-inflammatory (steroids or NSAIDs) or cough/cold or allergy preparation in the two weeks prior to the challenge

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 380 (Actual)
Dates: Start 2016-02; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turner RB, Lehtoranta L, Hibberd A, Mannikko S, Zabel B, Yeung N, Huttunen T, Burns FR, Lehtinen MJ. Effect of Bifidobacterium animalis spp. lactis Bl-04 on Rhinovirus-Induced Colds: A Randomized, Placebo-Controlled, Single-Center, Phase II Trial in Healthy Volunteers. EClinicalMedicine. 2021 Dec 3;43:101224. doi: 10.1016/j.eclinm.2021.101224. eCollection 2022 Jan. PMID 34927036

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All volunteers who signed consent were considered enrolled in the study per UVA IRB policy. 334 of these 380 volunteers were randomized to treatment after pre-treatment screening was complete.
Groups:
- Bifidobacterium Lactis Bl-04: 2*109 cfus of probiotic Bifidobacterium lactis Bl-04 (DuPont Nutrition and Health) mixed with 1g of sucrose as a carrier
  Bifidobacterium animalis subsp. lactis Bl-04
Period: Overall Study
Arm/Group | Bifidobacterium Lactis Bl-04 | Placebo
Started | 165 | 169
Completed | 143 | 153
Not Completed | 22 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bifidobacterium Lactis Bl-04 | Placebo | Total
Number analyzed (Participants) | 165 | 169 | 334
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.3 (6.7) | 22.2 (6.0) | 22.2 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 94 | 200
  Male | 59 | 75 | 134
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 11 | 17
  Not Hispanic or Latino | 132 | 130 | 262
  Unknown or Not Reported | 27 | 28 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 16 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 12 | 22
  White | 123 | 120 | 243
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 15 | 18 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Rhinovirus-associated Illness Episodes
Description: Rhinovirus-associated illness episodes: Volunteers who have both a rhinovirus infection and a symptomatic illness will be defined as having a rhinovirus-associated common cold illness.
Time Frame: 5 days
Population: Volunteers who were challenged with rhinovirus, completed the study period and did not have any evidence by PCR or serology of a viral infection with a virus other than the challenge virus
Measure: Count of Participants; unit: Participants
Arm/Group | Bifidobacterium Lactis Bl-04 | Placebo
Number analyzed (Participants) | 112 | 120
Participants | 63 | 60

ADVERSE EVENTS:
Time Frame: Consent/screening through the final study visit on study day 21-28.
Description: For the purposes of this study using experimental rhinovirus infection, physical signs and symptoms that are expected to be associated with the common cold should not be reported as adverse events. The following physical signs and symptoms are expected to be associated with the common cold: nasal obstruction (nasal stuffiness), coryza (runny nose), sore throat, cough, sneezing, myalgia, headache, feverishness, chills, loss of appetite and malaise.
Arm/Group | Bifidobacterium Lactis Bl-04 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/165 | 0/169
Serious Adverse Events (participants affected / at risk) | 1/165 | 0/169
Other Adverse Events (participants affected / at risk) | 89/165 | 84/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bifidobacterium Lactis Bl-04 (N=165) | Placebo (N=169)
achillles tendon rupture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bifidobacterium Lactis Bl-04 (N=165) | Placebo (N=169)
headache (General disorders) | 39 (51) | 35 (38)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 21 (21)
oropharyngeal pain (Gastrointestinal disorders) | 12 (15) | 15 (15)
cough (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 6 (6)
dysmenorrhea (Reproductive system and breast disorders) | 10 (13) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-13): https://cdn.clinicaltrials.gov/large-docs/07/NCT02679807/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/07/NCT02679807/SAP_001.pdf